CLINICAL TRIAL: NCT00498654
Title: A Randomized, Double-Blind, Multi-Center, Placebo-Controlled Dose Ranging Study to Determine the Safety, Reactogenicity and Immunogenicity of a Single Oral Dose Typhoid Fever Vaccine (Ty800) in Healthy Adult Subjects
Brief Title: Dose Ranging Study to Determine the Safety, Reactogenicity and Immunogenicity of Typhoid Fever Vaccine (Ty800) in Healthy Adult Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Avant Immunotherapeutics (Industry)
Responsible Party: AVANT Immnunotherapeutics
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Ty800-07-0001
Record Dates: First submitted 2007-07-09; First posted 2007-07-10 (Estimated); Last update posted 2008-07-02 (Estimated); Status verified 2008-06

CONDITIONS: Typhoid Fever
Keywords: Prevention of Typhoid Fever in Adult Travelers
MeSH Terms: conditions — Typhoid Fever | interventions — Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: Ty800 (Salmonella typhi) Oral Vaccine

SUMMARY:
The purpose of this trial is to examine the safety and immunogenicity of Ty800 oral vaccine in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Males or Females aged 18 to 55 years, inclusive
* Capable of understanding and complying with the protocol requirements and be available for the duration of the protocol

Exclusion Criteria:

* History of malignancy, immunocompromised conditions or currently receiving immunosuppressive treatment including systemic steroids
* History of Typhoid Fever infection, vaccination against typhoid fever or participation in a Clinical Trial using S.typhi organism at any time
* History of travel to a typhoid endemic region within the last 5 years or history of raising a child from an endemic area. Endemic regions are South and East Asia, the Indian Subcontinent, Africa and Central and South America including Mexico
* History of persistent diarrhea, blood in stool, peptic ulcer disease, or inflammatory bowel disease
* Allergies or sensitivities to antibiotics, notably quinolones, penicillins, sulfonamides, cefalosporins and chloramphenicol, and components of the buffer solution, notably aspartame.
* People who are commercial food handlers, day care workers, or health care workers involved in direct patient care. Also people with young children under 2 years of age at home or household contacts who are immunocompromised, pregnant or breast-feeding

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2007-07; Primary Completion 2007-10 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Immunogenicity | Baseline through Day 14
Reactogenicity | Baseline through Month 1 follow-up

SECONDARY OUTCOMES:
Longterm safety and immunogenicity | Month 1 to 6 post-dosing

CONTACTS AND LOCATIONS:
Overall Officials: Clark McKeever, MD, Principal Investigator — Accelovance LLC
Locations (5):
- United States (5):
  - Accelovance LLC, San Diego, California
  - Accelovance LLC, Melbourne, Florida
  - Accelovance LLC, Peoria, Illinois
  - Accelovance LLC, South Bend, Indiana
  - Accelovance LLC, Houston, Texas